CLINICAL TRIAL: NCT04524910
Title: A REtrospective Non-interventional Study to Assess the Effectiveness of AfLibercept in Patients With Myopic CNV
Brief Title: A Study to Learn More About How Drug Aflibercept Works in Canadian Patients With Reduced Vision Caused by New Blood Vessels Growing in the Eye (Myopic Choroidal Neovascularization or mCNV)
Acronym: REALM
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 20196
Record Dates: First submitted 2020-08-21; First posted 2020-08-24 (Actual); Last update posted 2023-06-18 (Actual); Status verified 2023-06

CONDITIONS: Myopic Choroidal Neovascularization
Keywords: Intravitreal Aflibercept; Choroidal Neovascularization; Vascular Endothelial Growth Factor (VEGF)
MeSH Terms: conditions — Choroidal Neovascularization | interventions — aflibercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- mCNV patients: Adult Canadian patients diagnosed with myopic choroidal neovascularization (mCNV) and naïve for anti-VEGF treatment
  Interventions: Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321)

INTERVENTIONS:
Drug: Aflibercept (Eylea, VEGF Trap-Eye, BAY86-5321) — As prescribed by the treating physician

SUMMARY:
Being short sighted means that vision is blurry when looking at things far away. People with a condition called "pathologic myopia" are short sighted due to problems in the back layer of their eyes, also known as the retina. Some people with pathologic myopia can develop a serious condition called myopic choroidal neovascularization (mCNV). In people with mCNV, new blood vessels grow into the retina. These blood vessels can break, leaking blood or fluid into the retina. This can cause blurry vision or a loss of vision.

In this study, researchers will find out more about how well drug aflibercept works and how safe it is in Canadian patients with mCNV.

The researchers in this study will review information from the patients' eye doctor visits. The patients in this study will include Canadian men and women who started receiving aflibercept between May 2017 and August 2019. These patients were at least 18 years old and had not received treatment for their mCNV before.

The researchers will look at the results of vision tests to find out how well the patients could read from a distance after they received aflibercept for 6 months. They will compare the results of these tests to before the patients received treatment. They will also learn more about how safe it is to have aflibercept injection into the eye.

ELIGIBILITY:
Inclusion Criteria:

* Adult (Age ≥ 18 years) female or male patient.
* Anti-VEGF treatment naïve patients diagnosed with mCNV.
* Initiation of treatment with aflibercept was made as per investigator's routine treatment practice between 01 MAY 2017 and 31 AUG 2019.

Exclusion Criteria:

* Any participation in an investigational program with interventions outside of routine clinical practice.
* Patients who have previously been treated with anti-VEGF intravitreal injections, systemic anti-VEGF or pro-VEGF treatments, as well as other intravitreal steroids or steroid implants for the study eye.
* Patients with another retinal disease (e.g. wet age-related macular degeneration,-wAMD; diabetic macular edema-DME; retinal vein occlusion-RVO), patients with advanced cataracts or glaucoma, or patients with scarring, fibrosis, or atrophy involving the center of the fovea.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients to be enrolled into the study must have been diagnosed with mCNV and started anti-VEGF treatment with aflibercept.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-11-11 (Actual)

PRIMARY OUTCOMES:
Change in best corrected visual acuity (BCVA) from baseline to 6 months | Baseline to 6 months
  BCVA is assessed by ETDRS (Early Treatment Diabetic Retinopathy Study) or Snellen chart with conversion to ETDRS.

SECONDARY OUTCOMES:
Change in BCVA from baseline to 12 months | Baseline to 12 months
  BCVA is assessed by ETDRS (Early Treatment Diabetic Retinopathy Study) or Snellen chart with conversion to ETDRS.
Central retinal thickness (in μm) measured by Optical coherence tomography (OCT) | At baseline, 6 and 12 months
  Retinal and lesion characteristics were evaluated using spectral domain optical coherence tomography (OCT).
Number of treatment-emergent adverse events (TEAS's) | Baseline to 12 months
  TEAEs comprise both ocular and non-ocular TEAEs
Severity of treatment-emergent adverse events | Baseline to 12 months
  TEAEs comprise both ocular and non-ocular TEAEs
Time from diagnosis to first treatment | At 12 months
Number of aflibercept treatments | At 12 months
Number of clinic visits | At 12 months
Number of visual acuity tests performed | At 12 months
Number of imaging assessments performed | At 12 months
Type of imaging assessments performed | At 12 months
  Imaging assessments as : OCT- Optical coherence tomography; OCTA- Optical coherence tomography angiography; FA- Fluorescein angiography and ICGA- Indocyanine green angiography

CONTACTS AND LOCATIONS:
Locations (1):
- Many Locations, Multiple Locations, Canada

IPD SHARING:
Plan to Share IPD: No
Availability of this study's data will later be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014.
  Interested researchers can use www.vivli.org to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the member section of the portal.